CLINICAL TRIAL: NCT03218046
Title: Eye Movement Desensitisation and Reprocessing (EMDR) as a Treatment for Tinnitus: A Feasibility Study
Brief Title: EMDR as a Treatment for Tinnitus
Acronym: EMDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julie Dawson (Other)
Responsible Party: Sponsor-Investigator, Julie Dawson, Research Services Manager, Norfolk and Norwich University Hospitals NHS Foundation Trust
Organization: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 174629
Record Dates: First submitted 2016-12-20; First posted 2017-07-14 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EMDR group (Experimental): This is the treatment arm that will receive EMDR therapy
  Interventions: Behavioral: EMDR

INTERVENTIONS:
Behavioral: EMDR — Eye Movement Desensitisation and Reprocessing

SUMMARY:
Tinnitus may be considered as a form of phantom auditory sensation and as such parallels may be drawn with other forms of phantom sensation, such as the sensation of pain in an amputated limb (phantom limb pain). There has been recent interest in the use of eye movement therapies to treat patients with phantom sensations such as these. The role of eye movements in the propagation and maintenance of tinnitus has also been well established. The main aim of this study is to evaluate the effectiveness of an established form of eye movement therapy called Eye Movement Desensitisation and Reprocessing (EMDR). This research is important as EMDR has produced encouraging results for other forms of phantom sensation and current models of tinnitus fit well with the proposed mode of action of EMDR. Tinnitus is very prevalent in our population and is often associated with significant discomfort; however, there is a severe lack of effective treatments based on well designed clinical trials. The investigator wishes to assess the usefulness of EMDR against the current treatment that is available in many institutions including the Investigator's own. The Investigator intends to recruit 15-30 patients initially to run a pilot study, before embarking on a larger scale study. The Investigator hopes that this pilot study will run over the course of a year. If this study demonstrates a significant improvement in tinnitus in patient undergoing EMDR, this will be an important step forward not only for treating patients with this disorder, but also for understanding the pathways that initiate, propagate and maintain tinnitus perception.

DETAILED DESCRIPTION:
Tinnitus is a common, yet poorly understood condition. In the UK, a large study using data from more than 500,000 people has found a prevalence of tinnitus of 16.2% (defined as any noise in the ear/s lasting longer than five minutes) and a prevalence of bothersome tinnitus as 3.8% (those who were moderately or severely bothered by their tinnitus on a four point Likert scale). Other international studies have also found a high prevalence of 30% with a total of 6% of the study population reporting incapacitating symptoms from tinnitus. Despite the high worldwide prevalence of tinnitus and the large number of proposed therapies available, there is a distinct paucity of well controlled trials in the literature to support an effective treatment.

Tinnitus may be considered as a form of phantom auditory perception and as such parallels may be drawn with other forms of phantom sensation, there has been recent interest in the use of eye movement therapies to treat patients with phantom sensations such as phantom limb pain. Both studies of those with tinnitus and phantom limb pain have suggested a psychological component such as certain premorbid personality traits may also contribute or predispose to these conditions and consequently be helped by psychological therapies.

Eye Movement Desensitisation and Reprocessing (EMDR) was first described by Shapiro in 1989 and requires the subject to perform relatively rapid movements of the eyes. Its application has been particularly documented in the context of post-traumatic stress disorder (PTSD). EMDR has been described as an integrative psychotherapy, due to its assimilation of various elements from diverse psychotherapies. A number of models have been proposed to account for the role of eye movements in EMDR, these include Shapiro's Adaptive Information Processing Model, Dyck's conditioning model, attentional processing accounts and theories of reverse learning . A recurrent mechanism in a number of these accounts is that of the orientating reflex. MacCollock and Feldman argue that lateral eye-movements trigger an investigatory component of this reflex to assess safety with regard to potential external threats . Where threats are positively identified, a flight or flight response is initiated; in situations where no danger is identified a functional reduction in arousal takes place. Support for this reassurance response in non-clinical patients has been demonstrated using auditory stimuli. Overlap between these concepts and theories related to the perception of tinnitus bode well, especially when one considers the neurophysiological model proposed by Jastreboff.

Since its introduction in 1989, numerous controlled studies have been conducted to evaluate EMDR's utility as a treatment for various forms of trauma-related complaints, including PTSD. The positive results have established EMDR as an effective trauma treatment and have prompted numerous professional organisations to recognise its efficacy, beginning with the American Psychological Association's (APA) Division 12 Task Force on Psychological Interventions in 1998. Since then, the NHS the International Society for Traumatic Stress Studies , the Israeli National Council for Mental Health , and the Northern Ireland Department of Health have also supported EMDR. Most recently, the US Departments of Defence and Veterans Affairs stated that EMDR was an effective treatment of trauma, as did the American Psychiatric Association . It has also been found to be helpful in medically unexplained symptoms and somatoform disorders.

Other forms of eye movement therapy have been popularised, such as eye movement integration therapy (EMI) in which eye movements in specific directions provide access strategies to different sensory domains. EMI was originally developed from research in the field of neuro-linguistic programming (NLP) and has also been widely used in the treatment of PTSD. EMI uses slower eye movements that are thought to access internal dialogue or emotional and feeling areas of the brain. Initially the concept of specifically accessing domains associated with auditory-based cue was appealing as a therapy for an auditory based pathology, however, despite initial enthusiasm for EMI the specificity of these associations has been disputed.

The role of eye movements in the propagation and maintenance of tinnitus has been well established, although the exact neurophysiological mechanisms of how eye movements integrate within the central auditory areas is not fully understood, however functional imaging has suggested a number of neuroanatomical sites. Cognitive science has provided neural networks that model tinnitus, these neural network models were inspired by theoretical models that described possible neural mechanisms mediating tinnitus. The majority of these models rely on the lateral-inhibition network (LIN) to simulate tinnitus and focus on the role of central auditory processing regions as possible anatomical locations of the physiological abnormalities that cause tinnitus. Recent work has identified a number of regions responsible for the generation and modulation of tinnitus including limbic, somatosensory and motor areas.

There has been some encouraging work described in the German literature regarding the effectiveness of EMDR for the treatment of tinnitus. The application of eye movement therapies to treat patients with tinnitus would seem logical considering the context our current understanding of tinnitus; the next step would be to test this theory in the setting of a formal randomised controlled clinical study.

ELIGIBILITY:
Inclusion Criteria:

- 1. 'Subjective Idiopathic Tinnitus', specifically 'Chronic Decompensated Tinnitus' with a THI score of 38 to 100.

2. Tinnitus for greater than 6 months duration. 3. Aged over 18 4. Willing to commit to a full course of EMDR therapy

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Change in tinnitus handicap inventory score | 6 months
  Tinnitus questionnaire

SECONDARY OUTCOMES:
Beck Depression Inventory (T0, T1, T2) | 6 months
  Depression questionnaire
Beck Anxiety Inventory(T0, T1, T2) | 6 months
  Anxiety questionnaire
Posttraumatic Stress Diagnostic Scale (T0, T1, T2) | 6 months
  Post traumatic stress questionnaire
Pure Tone Audiogram (T0). | 6 months
  Hearing test
Psychoacoustic parameters: (T0, T1, T2) a. Intensity - Tinnitus loudness estimate using a VAS b. Loudness Discomfort Level (LDL) at 250-8000Hz | 6 months
  Quasi objective measure of tinnitus
Five factor personality inventory (T0) | 6 months
  Personality questionnaire
Free text evaluation of treatment and trial protocol (T2) | 6 months
  Open appraisal of study

CONTACTS AND LOCATIONS:
Overall Officials: John Phillips, Principal Investigator — Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK)
Locations (1):
- Norfolk and Norwich University Hospital, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Background] Lockwood AH, Salvi RJ, Burkard RF. Tinnitus. N Engl J Med. 2002 Sep 19;347(12):904-10. doi: 10.1056/NEJMra013395. No abstract available. PMID 12239260
- [Background] Noell CA, Meyerhoff WL. Tinnitus. Diagnosis and treatment of this elusive symptom. Geriatrics. 2003 Feb;58(2):28-34. PMID 12596495
- [Background] Davis A, El Rafaie A. Epidemiology of tinnitus. In: Tyler RS, (ed). Tinnitus Handbook. San Diego: Singular, 2000; 1-23.
- [Background] McFerran DJ, Phillips JS. Tinnitus. J Laryngol Otol. 2007 Mar;121(3):201-8. doi: 10.1017/S0022215106002714. Epub 2006 Sep 25. PMID 16995967
- [Background] Oren, E. and R. Solomon (2012).
- [Background] Flor H. Phantom-limb pain: characteristics, causes, and treatment. Lancet Neurol. 2002 Jul;1(3):182-9. doi: 10.1016/s1474-4422(02)00074-1. PMID 12849487
- [Background] Shapiro F. Efficacy of the eye movement desensitization procedure in the treatment of traumatic memories. J Trauma Stress. 1989;2(2):199-223.
- [Background] Bisson J, Andrew M. Psychological treatment of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2007 Jul 18;(3):CD003388. doi: 10.1002/14651858.CD003388.pub3. PMID 17636720
- [Background] Shapiro F. Eye Movement Desensitization and Reprocessing (EMDR): Basic Principles, Protocols, and Procedures, 2nd Edition. 2001. The Guilford Press.
- [Background] Dyck MJ. A proposal for a conditioning model of eye movement desensitization treatment for posttraumatic stress disorder. J Behav Ther Exp Psychiatry. 1993 Sep;24(3):201-10. doi: 10.1016/0005-7916(93)90022-o. PMID 7910613
- [Background] Kuiken D, Bears M, Miall D, Smith L. Eye Movement Desensitisation Reprocessing Facilitates Attentional Orienting. Imagination, Cognition and Personality. 2002;21:3-20.
- [Background] Hassard A. Reverse learning and the physiological basis of eye movement desensitization. Med Hypotheses. 1996 Oct;47(4):277-82. doi: 10.1016/s0306-9877(96)90067-5. PMID 8910876
- [Background] MacCulloch MJ, Feldman P. Eye movement desensitisation treatment utilises the positive visceral element of the investigatory reflex to inhibit the memories of post-traumatic stress disorder: a theoretical analysis. Br J Psychiatry. 1996 Nov;169(5):571-9. doi: 10.1192/bjp.169.5.571. PMID 8932885
- [Background] Barrowcliff AL, Gray NS, MacCulloch S, Freeman TC, MacCulloch MJ. Horizontal rhythmical eye movements consistently diminish the arousal provoked by auditory stimuli. Br J Clin Psychol. 2003 Sep;42(Pt 3):289-302. doi: 10.1348/01446650360703393. PMID 14565894
- [Background] Jastreboff PJ. Phantom auditory perception (tinnitus): mechanisms of generation and perception. Neurosci Res. 1990 Aug;8(4):221-54. doi: 10.1016/0168-0102(90)90031-9. PMID 2175858
- [Background] National Institute for Clinical Excellence (2005). Post traumatic stress disorder (PTSD): The management of adults and children in primary and secondary care. London: NICE Guidelines. . http://www.oqp.med.va.gov/cpg/PTSD/PTSD_cpg/frameset.htm
- [Background] Ursano RJ, Bell C, Eth S, Friedman M, Norwood A, Pfefferbaum B, Pynoos JD, Zatzick DF, Benedek DM, McIntyre JS, Charles SC, Altshuler K, Cook I, Cross CD, Mellman L, Moench LA, Norquist G, Twemlow SW, Woods S, Yager J; Work Group on ASD and PTSD; Steering Committee on Practice Guidelines. Practice guideline for the treatment of patients with acute stress disorder and posttraumatic stress disorder. Am J Psychiatry. 2004 Nov;161(11 Suppl):3-31. No abstract available. PMID 15617511
- [Background] van Rood, Y. R. and C. de Roos (2009).
- [Background] Farmer A, Rooney R, Cunningham JR. Hypothesized eye movements of neurolinguistic programming: a statistical artifact. Percept Mot Skills. 1985 Dec;61(3 Pt 1):717-8. doi: 10.2466/pms.1985.61.3.717. PMID 4088761
- [Background] Wertheim EH, Habib C, Cumming G. Test of the neurolinguistic programming hypothesis that eye-movements relate to processing imagery. Percept Mot Skills. 1986 Apr;62(2):523-9. doi: 10.2466/pms.1986.62.2.523. PMID 3503261
- [Background] Baguley DM, Phillips J, Humphriss RL, Jones S, Axon PR, Moffat DA. The prevalence and onset of gaze modulation of tinnitus and increased sensitivity to noise after translabyrinthine vestibular schwannoma excision. Otol Neurotol. 2006 Feb;27(2):220-4. doi: 10.1097/01.mao.0000172412.87778.28. PMID 16436993
- [Background] Coad ML, Lockwood A, Salvi R, Burkard R. Characteristics of patients with gaze-evoked tinnitus. Otol Neurotol. 2001 Sep;22(5):650-4. doi: 10.1097/00129492-200109000-00016. PMID 11568674
- [Background] Biggs ND, Ramsden RT. Gaze-evoked tinnitus following acoustic neuroma resection: a de-afferentation plasticity phenomenon? Clin Otolaryngol Allied Sci. 2002 Oct;27(5):338-43. doi: 10.1046/j.1365-2273.2002.00591.x. PMID 12383293
- [Background] Lockwood AH, Wack DS, Burkard RF, Coad ML, Reyes SA, Arnold SA, Salvi RJ. The functional anatomy of gaze-evoked tinnitus and sustained lateral gaze. Neurology. 2001 Feb 27;56(4):472-80. doi: 10.1212/wnl.56.4.472. PMID 11222790
- [Background] Husain FT. Neural network models of tinnitus. Prog Brain Res. 2007;166:125-40. doi: 10.1016/S0079-6123(07)66011-7. PMID 17956777
- [Background] Moller AR. Pathophysiology of tinnitus. Ann Otol Rhinol Laryngol. 1984 Jan-Feb;93(1 Pt 1):39-44. PMID 6367601